CLINICAL TRIAL: NCT00508521
Title: Treatment of Hand Dysfunction After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B4078-R
Record Dates: First submitted 2007-07-27; First posted 2007-07-30 (Estimated); Results first posted 2014-02-07 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2013-12

CONDITIONS: Stroke
Keywords: cerebrovascular accident; electrical stimulation; motor learning; upper extremity rehabilitation
MeSH Terms: conditions — Stroke | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FES and Motor Learning Training (Experimental): participants <6 months after first stroke who presented with arm dysfunction were trained using FES and Motor Learning
  Interventions: Device: Functional Electrical Stimulation
- Control group (Other): Subjects in this arm will receive standard care as prescribed by their physician and covered by their insurance
  Interventions: Other: Standard Care

INTERVENTIONS:
Device: Functional Electrical Stimulation — commercially available surface electrical stimulator
  Arms: FES and Motor Learning Training
Other: Standard Care — Standard care as ordered by their physician and covered by their insurance company.
  Arms: Control group

SUMMARY:
Many stroke survivors exhibit persistent upper limb motor deficits and a non-functional upper limb. There is some promising information that suggests motor learning (ML) in conjunction with functional electrical stimulation (FES; surface FES; nothing implanted; use of a commercially available system) of wrist/finger muscles can significantly enhance the functional level of the upper limb. There have been promising studies showing that some subjects in the chronic phase (greater than 6 months after stroke) responded favorably to combination FES and ML (FES ML). In our pilot studies, FES ML for those in the chronic phase (>12 months) produced statistically significant functional recovery. FES was applied using a commercially available, two-channel FES system, with electrodes applied to the surface of the skin (non-invasive). But if upper limb dysfunction is not immediately treated, that is within the sub-acute phase (less than 6 months) following stroke, the following problems can develop: contractures and other soft tissue changes; chronic pain; and ingrained, abnormal, non-functional movement patterns. The more long-standing these symptoms are, the more resistant to treatment they become. Therefore, it is important to provide promising interventions prior to the onset of chronic symptoms and dysfunction. Those in the sub-acute phase after stroke should be provided with FES ML, in order to more completely restore function for a greater number of stroke survivors.

Specific Aims and Hypotheses The goal of this pilot study is to test the feasibility of the proposed treatment in the sub acute phase following stroke.

HYPOTHESIS. FES ML for 3hrs/day, five days/week, for 12 weeks will be feasible to implement in the sub-acute phase following stroke (2 -24 weeks).

Study Design

a. Specific Procedures This is a pilot study to test the feasibility of using FES ML for upper extremity rehabilitation in a sub-acute stroke population. It is a randomized, controlled, single-blind design. Subjects will be 2 - 24 weeks after a single stroke. The control group will receive standard care for upper limb rehabilitation consisting of passive and active exercise, stretching, bracing, and use of adaptive devices. The experimental group will receive the experimental intervention in addition to their standard care.

CONTROL GROUP INTERVENTION. The control group will receive the standard medical care prescribed by the primary physician and covered by the subject's health care policy. Standard care will include: soft tissue mobilization; assisted motion exercise; active motion exercise; resistive exercise; task practice; use of assistive devices; and modality applications conventionally prescribed.

FES ML INTERVENTION. The research treatment duration will be 3hrs/day, five days per week. The subjects will be present for a fourth hour each day, which will be used for breaks and rest periods that will be interspersed throughout the intervention time. The treatment duration is derived from prior work. We will stimulate muscles in a number of configurations including: wrist extension and finger extension; wrist extension and finger flexion; and wrist extension, finger flexion, and thumb abduction and opposition. Motor learning will include the performance of functional task components and full task practice during the use of FES. FES will be triggered by the patient, the treating therapist, or it will be automatically sequenced by the device according to alternate channel activations, with timings pre-set by the treating therapist.

MEASURES. Data will be collected at weeks 1, 6, 12 (end of treatment), and 6 months after the end of treatment.

Population The subjects will be sub-acute stroke survivors (2-24 weeks after stroke).

ELIGIBILITY:
Inclusion Criteria:

* 2-24 weeks after stroke
* Greater than 21 years old
* Ability to follow 2 step commands

Exclusion Criteria:

* Chronic, progressive medical condition (i.e. Parkinson's Disease)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-01; Primary Completion 2010-01 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janis Daly, PhD MS, Principal Investigator — VA Medical Center-Cleveland
Locations (1):
- VA Medical Center, Cleveland, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited through the use of study flier and by word of mouth.
Pre-assignment Details: All subjects enrolled in the study were entered into the same arm of this pilot study
Groups:
- FES and Motor Learning Training Group: Subjects < 6 months following first stroke who had diminished upper limb strength, coordination and function.
Period: Overall Study
Arm/Group | FES and Motor Learning Training Group
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1 Subjects With Acute Stroke: Subjects < 6 months following first stroke who had diminished upper limb strength, coordination and function.
Arm/Group | Arm 1 Subjects With Acute Stroke
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Fugl-Meyer Upper Limb Coordination Scale (FMUE)
Description: A subscale of the Fugl-Meyer; the Fugl-Meyer Upper Limb Coordination Scale is a measure of movement coordination in and out of synergy patterns for the hemiparetic upper limb; scores range from 0-66, with 0 being the worst score and 66 being the best score.
Time Frame: baseline and after 12 weeks of training
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 Subjects With Acute Stroke
Number analyzed (Participants) | 4
units on a scale
  Pre-Treatment Fugl Meyer Upper Limb Score | 27.75 (3.86)
  Post-Treatment Fugl Meyer Upper Limb Score | 48.50 (3.16)
Statistical Analysis 1: Comparison: Arm 1 Subjects With Acute Stroke; This was a feasibility study. Pre and post treatment analysis was performed for the study participants; Test type: Superiority or Other; p = .0001, t-test, 2 sided; Mean Difference (Final Values) = -20.75, 95% CI 2-sided [-22.27348 to -19.22652], Standard Error of Mean .47871

ADVERSE EVENTS:
Arm/Group | Arm 1 Subjects With Acute Stroke
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
This was a small pilot feasibility study providing data for future work.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes